CLINICAL TRIAL: NCT06076096
Title: Ultrasound-Guided Supra-Inguinal Fascia Iliaca Block As an Anesthesia Method for Lower Extremity Surgeries: A Single-Center Retrospective Cohort Feasibility Study
Brief Title: SIFIB As an Anesthesia Method for Lower Extremity Surgeries
Status: Completed | Type: Observational
Sponsor: Samsun University (Other)
Responsible Party: Sponsor
Other Study IDs: SIFIB retrospective
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Anesthesia; Anesthesia Management; Regional Anesthesia
Keywords: Regional Anesthesia; Anesthesia Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Suprainguinal fascia iliaca block — The design of this study involved the retrospective analysis of data. Data was gathered from adult patients falling into the American Society of Anesthesiology (ASA) categories I to III, who were scheduled for elective lower limb surgical procedures. More specifically, patients who had undergone SIFIB either as the primary anesthesia approach or as part of their anesthesia regimen were included. Those who had received general anesthesia, neuraxial anesthesia, or infiltration anesthesia were excluded from the study. Importantly, all patients who participated in the study provided written informed consent for both their involvement in the study and the publication of their data.
  Other Names: Sciatic nerve block

SUMMARY:
The Ultrasound-guided Supra-inguinal Fascia Iliaca Block (SIFIB) is an advanced regional anesthesia technique strategically directed at the three primary nerves of the lumbar plexus. As the scope of regional anesthesia methods continues to grow in clinical application, this approach emerges as a versatile method. It can be used independently for pain management or as the primary anesthetic method, particularly in well-selected patients undergoing isolated limb surgeries or in combination with other regional anesthesia approaches.

DETAILED DESCRIPTION:
The study follows a retrospective cohort feasibility design, conducted within the confines of a tertiary hospital. The requisite data for analysis was acquired by accessing patient records and electronic data systems. A cohort of 16 patients was carefully chosen for inclusion in the study, and the administration of blocks was carried out before the surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients who underwent elective lower limb surgical procedures.

Exclusion Criteria:

* Patients who received general anesthesia, neuraxial anesthesia, or infiltration anesthesia were excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Specifically, we included patients who underwent SIFIB either as the primary anesthesia method or as a component of the anesthesia plan.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Block Success which provided surgical anesthesia, intraoperatively | Intraoperatively and PACU unit (up to 2 hours)
  After performing the blocks, the sensory block was examined with a pinprick test using a 27-gauge hypodermic needle, (0 = no sensory block; 1 = tactile sense present, no pain; 2 = no tactile sense and no pain). Cases with a score of 1 or 2 after 30 min were considered successful.

SECONDARY OUTCOMES:
Additional analgesic requirement | Intraoperatively and PACU unit (up to 2 hours)
  The number of patient who required intravenous ketamine or propofol infusion were recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Serkan Tulgar, M.D., Study Director — Samsun University
Locations (1):
- Samsun University, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided